CLINICAL TRIAL: NCT06191328
Title: A Prospective, Open, Self-controlled Study of the Effects of Chiglitazar Sodium on Glucose and Lipid Metabolism in Patients With Type 2 Diabetes Mellitus (T2DM)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yufan Wang (Other)
Responsible Party: Sponsor-Investigator, Yufan Wang, Professor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CGZIIT013
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental)
  Interventions: Drug: Chiglitazar sodium

INTERVENTIONS:
Drug: Chiglitazar sodium — In patients with type 2 diabetes mellitus (T2DM), on the basis of one or two oral hypoglycemic agents combination with Chiglitazar sodium.

SUMMARY:
The goal of this clinical trial is to learn about inour study aimed to evaluate serum lipid profiles of T2DM patients before and after Chiglitazar Sodium administration.

The main question[s] it aims to answer are:

* Quantitative lipidomics information enables in-depth analysis of lipids and can reveal Chiglitazar Sodium-specific lipid metabolic patterns, thereby strengthening lipidomics as a promising tool for exploring the molecular mechanisms of T2DM.
* It can also be applied to other T2DM lipidomics studies to better understand lipid metabolism patterns and integration with other omics measures.

DETAILED DESCRIPTION:
Chiglitazar Sodium for lipid profile abnormalities and its associated effective lipid molecular biomarkers have never been studied in patients with T2DM. Therefore, our study aimed to evaluate serum lipid profiles of T2DM patients before and after Chiglitazar Sodium administration using ultra-high performance liquid chromatography-Tandem quadrupole time-of-flight mass spectrometry (UPLC-QTOF-MS). For completeness, we also evaluated the effects of Chiglitazar Sodium treatment on metabolic markers associated with T2DM and its association with lipidomic changes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with type 2 diabetes (T2DM) WHO meet the diagnostic criteria for diabetes issued by the World Health Organization (WHO) in 1999;
2. Male or female patients aged ≥18, ≤70 years;
3. BMI≥18.5 Kg/m2, < 35 Kg/m2;
4. Hemoglobin a1C (HbA1C) ≥7.5%; ≤10.5%;
5. Triglyceride ≤500 mg /dL (5.65 mmol/L) (if the researchers judge that the transient increase caused by diet, etc., can be repeated detection)
6. Total cholesterol (TC) ≤250mg/dl (6.45mmol/L)
7. T2DM patients who are taking one or two kinds of oral hypoglycemic drugs with fixed dose ≥2 months and uncontrolled blood glucose.
8. Voluntarily sign informed consent and agree to enter the trial group.

Exclusion Criteria:

1. Type 1 diabetes or other specific type of diabetes
2. Fasting blood glucose (FPG) > 13.3 mmol/L (240 mg/dL);
3. Triglyceride (TG) > 500 mg /dL (5.65 mmol/L);
4. Total cholesterol (TC) > 250mg/dl (> 6.45mmol/L);
5. Refractory hypertension [that is, on the basis of improving the lifestyle, the blood pressure is still not up to standard after 1 month of applying a reasonably tolerable amount of 3 or more antihypertensive drugs (including diuretics), or the blood pressure can be effectively controlled by taking 4 or more antihypertensive drugs;
6. Taking fibrates, statins, thiazolidinediones, insulin drugs;
7. A clear diagnosis of severe osteoporosis or any other known bone disease;
8. A history of diabetic ketoacidosis, diabetic hyperglycemia hyperosmolar syndrome, lactic acidosis and other acute complications of diabetes;
9. Severe microvascular complications (proliferative retinopathy; Urinary albumin/creatinine ratio > 300 mg/g; Marked peripheral neuropathy, etc.);
10. The New York Heart Association (NYHA) defines congestive heart failure as grade III or IV;
11. Significant liver and kidney dysfunction and systemic disease (significant liver dysfunction is defined as AST> 2.5 times the upper limit of normal and/or ALT> 2.5 times the upper limit of normal and/or total bilirubin > 1.5 times the upper limit of normal value; Renal dysfunction was defined as moderate to severe renal insufficiency (eGFR<60 ml/ (min*1.73m2));
12. Pregnant or lactating women, women of childbearing age who are unable or unwilling to take adequate contraception;
13. Participating in a clinical trial of another drug or medical device in or within 3 months prior to screening;
14. The investigator considers it inappropriate to participate in this clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-31 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 12 weeks of treatment
  Change in HbA1c from baseline

SECONDARY OUTCOMES:
Serum lipid profile | 12 weeks of treatment
  Changes from baseline in sphingomyelin (SMs), ceramide (CER), lysophosphatidylcholine (LPC), phosphatidylethanolamine (PEs), lysophosphatidylethanolamine (LPEs), and phosphatidylcholine (PC)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai First People's Hospital, Shanghai, Shanghai Municipality, China